CLINICAL TRIAL: NCT00640224
Title: Obesity, Insulin Resistance, and Bone Metabolism in Adolescents With PCOS: Effects of Insulin Sensitizers Versus Oral Contraceptives
Brief Title: Insulin Resistance, Polycystic Ovary Syndrome, and Bone Research Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Silva Arslanian (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Silva Arslanian, Principal Investigator, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0503013; 2K24HD001357 (NIH)
Record Dates: First submitted 2008-03-18; First posted 2008-03-21 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-10

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Rosiglitazone; drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Rosiglitazone (Active Comparator): Treatment naive overweight adolescent females with PCOS treated with Rosiglitazone
  Interventions: Drug: rosiglitazone
- Drospirenone/ethinyl estradiol (Active Comparator): Treatment naive overweight adolescent females with PCOS treated with Drospirenone/ethinyl estradiol
  Interventions: Drug: drospirenone/ethinyl estradiol
- Overweight/Obese without PCOS (No Intervention): Overweight adolescent females without PCOS to use as comparison of normal developmental changes. *No participants were enrolled in this Arm.
- Lean without PCOS (No Intervention): Lean healthy girls without PCOS to serve as controls for the cardiovascular markers. *No participants were enrolled in this Arm.

INTERVENTIONS:
Drug: rosiglitazone — 4 mg daily for 6 months
  Other Names: Avandia
  Arms: Rosiglitazone
Drug: drospirenone/ethinyl estradiol — 1 tab (3mg/30mcg) daily for 6 months
  Other Names: Yasmin
  Arms: Drospirenone/ethinyl estradiol

SUMMARY:
The purpose is to investigate the effects of 2 different treatments (drospirenone/ethinyl estradiol versus rosiglitazone) on insulin sensitivity and androgen levels, inflammatory markers, vascular markers and bone development in overweight adolescent females with polycystic ovary syndrome (PCOS).

DETAILED DESCRIPTION:
The purpose of this study is to:

1) to compare effects of treatment with drospirenone/ethinyl estradiol (Yasmin)versus rosiglitazone (Avandia) on hyperandrogenism, insulin resistance/hyperinsulinemia, adrenal hyperresponsiveness, body composition, chronic inflammation, bone mass and turnover.

OCPs are the first-line therapy for PCOS, however, they do not address the insulin resistance or the inflammation. Insulin sensitizers have been used successfully to treat PCOS but thiazolidinediones such as rosiglitazone have not been used in adolescents. Therefore we will investigate the effects of treatment with drospirenone/ethinyl estradiol versus rosiglitazone in overweight adolescents with PCOS. We will obtain comprehensive evaluations before and 6 months after randomization, to the respective treatment arms to determine the differences between the 2 treatment modalities.

ELIGIBILITY:
Inclusion Criteria:

* Age 10 - 20 years
* Pubertal level of Tanner stage III-V and menarchal
* BMI percentile for age and sex greater than or equal to 85%ile

Exclusion Criteria:

* Oral medications for PCOS, or that have impact on bone (i.e. anti-epileptics)
* Presence of other diseases, systemic or psychiatric, or chronic medications which could interfere with endocrine function
* Established diagnosis of diabetes
* Prior bone surgery, prior osteoporotic fracture, or fracture in the past 12 months
* Prior thromboembolic event, such as a deep venous thrombosis or pulmonary embolism (PCOS subjects only)
* Vitamin D deficiency (<10ng/mL)
* Hyperkalemia (K>5.0 meq/L)
* Positive pregnancy test (serum)

Ages: 10 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 65 (Actual)
Dates: Start 2005-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Silva Arslanian, M.D., Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Tfayli H, Ulnach JW, Lee S, Sutton-Tyrrell K, Arslanian S. Drospirenone/ethinyl estradiol versus rosiglitazone treatment in overweight adolescents with polycystic ovary syndrome: comparison of metabolic, hormonal, and cardiovascular risk factors. J Clin Endocrinol Metab. 2011 May;96(5):1311-9. doi: 10.1210/jc.2010-2547. Epub 2011 Feb 16. PMID 21325466

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overweight/obese patients with PCOS were recruited from the Children's Hospital of Pittsburgh (CHP) PCOS center and the community through advertisements and flyers posted in the medical campus and in pediatricians' offices.
Pre-assignment Details: 9 did not meet diagnostic criteria, 3 were on psychiatric meds,1 was diagnosed with diabetes,1 had venous access issues, and 5 did not complete baseline evaluations. No participants were enrolled in the "Overweight/Obese without PCOS" or "Lean without PCOS" Arms/Groups.
Groups:
- Overweight/Obese Without PCOS: Overweight adolescent females without PCOS to use as comparison of normal developmental changes.
- Lean Without PCOS: Lean healthy girls without PCOS to serve as controls for the cardiovascular markers
Period: Overall Study
Arm/Group | Rosiglitazone | Drospirenone/Ethinyl Estradiol | Overweight/Obese Without PCOS | Lean Without PCOS
Started | 23 | 23 | 0 | 0
Completed | 17 | 20 | 0 | 0
Not Completed | 6 | 3 | 0 | 0
Not completed — Lost to Follow-up | 5 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Headaches | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rosiglitazone | Drospirenone/Ethinyl Estradiol | Overweight/Obese Without PCOS | Lean Without PCOS | Total
Number analyzed (Participants) | 17 | 20 | 0 | 0 | 37
Age, Categorical [Count of Participants; unit: Participants]
  Age: <=18 years | 16 | 18 |  |  | 34
  Age: Between 18 and 65 years | 1 | 2 |  |  | 3
  Age: >=65 years | 0 | 0 |  |  | 0
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 15.7 (4.1) | 16.2 (4.5) |  |  | 16.0 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 20 |  |  | 37
  Male | 0 | 0 |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 20 |  |  | 37

OUTCOME MEASURES:

1. Primary Outcome: Peripheral Insulin Sensitivity at Baseline and 6 Months.
Description: Peripheral insulin sensitivity was evaluated during the hyperinsulinemic-euglycemic clamp.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: mg/kg/min per uU/mL
Arm/Group | Rosiglitazone | Drospirenone/Ethinyl Estradiol | Overweight/Obese Without PCOS | Lean Without PCOS
Number analyzed (Participants) | 17 | 20 | 0 | 0
mg/kg/min per uU/mL
  Peripheral insulin sensitivity, Baseline | 2.2 (0.2) | 2.1 (0.2) |  |
  Peripheral insulin sensitivity, 6 months | 3.2 (0.4) | 2.0 (0.2) |  |

2. Primary Outcome: Hepatic Insulin Sensitivity at Baseline and 6 Months.
Description: Hepatic insulin sensitivity was evaluated prior to the hyperinsulinemic-euglycemic clamp.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: (mg/kg/min x uU/mL)-1
Arm/Group | Rosiglitazone | Drospirenone/Ethinyl Estradiol | Overweight/Obese Without PCOS | Lean Without PCOS
Number analyzed (Participants) | 17 | 20 | 0 | 0
(mg/kg/min x uU/mL)-1
  Hepatic insulin sensitivity, Baseline | 17.3 (1.8) | 17.4 (2.2) |  |
  Hepatic insulin sensitivity, 6 months | 24.1 (3.4) | 16.8 (2.2) |  |

3. Primary Outcome: Glucose Tolerance Status at Baseline and 6 Months.
Description: Glucose tolerance status was classified according to the ADA (American Diabetes Association) criteria.
Time Frame: Baseline and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Rosiglitazone | Drospirenone/Ethinyl Estradiol | Overweight/Obese Without PCOS | Lean Without PCOS
Number analyzed (Participants) | 17 | 20 | 0 | 0
Participants
  Normal glucose tolerance, baseline | 15 | 12 |  |
  Impaired glucose tolerance, baseline | 2 | 8 |  |
  Normal glucose tolerance, 6 months | 15 | 13 |  |
  Impaired glucose tolerance, 6 months | 2 | 7 |  |

4. Secondary Outcome: Total Fat Mass at Baseline and 6 Months
Description: DXA (dual-energy x-ray absorptiometry) scans were done to measure total fat mass.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: Kg
Arm/Group | Rosiglitazone | Drospirenone/Ethinyl Estradiol | Overweight/Obese Without PCOS | Lean Without PCOS
Number analyzed (Participants) | 17 | 20 | 0 | 0
Kg
  Fat mass, Baseline | 44.5 (2.8) | 48.0 (3.2) |  |
  Fat mass, 6 months | 45.4 (3.4) | 49.1 (3.4) |  |

5. Secondary Outcome: Total Testosterone at Baseline and 6 Months
Description: Total testosterone was measured by HPLC(high-performance liquid chromatography)-tandem mass spectroscopy.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: ng/dL
Arm/Group | Rosiglitazone | Drospirenone/Ethinyl Estradiol | Overweight/Obese Without PCOS | Lean Without PCOS
Number analyzed (Participants) | 17 | 20 | 0 | 0
ng/dL
  Total Testosterone, Baseline | 45.7 (5.6) | 34.5 (3.2) |  |
  Total Testosterone, 6 months | 36.9 (3.7) | 30.6 (3.1) |  |

6. Secondary Outcome: Percent Body Fat at Baseline and 6 Months
Description: DXA scans were done to measure the percentage of body fat.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: percentage of body fat
Arm/Group | Rosiglitazone | Drospirenone/Ethinyl Estradiol | Overweight/Obese Without PCOS | Lean Without PCOS
Number analyzed (Participants) | 17 | 20 | 0 | 0
percentage of body fat
  Percent body fat, Baseline | 46.2 (1.1) | 47.3 (1.1) |  |
  Percent body fat, 6 months | 46.6 (1.6) | 48.2 (1.2) |  |

7. Secondary Outcome: Free Testosterone at Baseline and 6 Months
Description: Free testosterone was measured by equilibrium dialysis.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Rosiglitazone | Drospirenone/Ethinyl Estradiol | Overweight/Obese Without PCOS | Lean Without PCOS
Number analyzed (Participants) | 17 | 20 | 0 | 0
pg/mL
  Free Testosterone, Baseline | 10.7 (2.0) | 7.5 (0.9) |  |
  Free Testosterone, 6 months | 7.7 (1.6) | 1.9 (0.3) |  |

8. Secondary Outcome: SHBG at Baseline and 6 Months
Description: SHBG (sex hormone-binding globulin) was measured by immunoradiometric assay.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Rosiglitazone | Drospirenone/Ethinyl Estradiol | Overweight/Obese Without PCOS | Lean Without PCOS
Number analyzed (Participants) | 17 | 20 | 0 | 0
nmol/L
  SHBG, Baseline | 28.1 (4.6) | 22.7 (2.2) |  |
  SHBG, 6 months | 37.0 (6.6) | 154.5 (24.0) |  |

9. Secondary Outcome: DHEAS at Baseline and 6 Months
Description: DHEAS (dehydroepiandrosterone sulfate) was measured by radioimmunoassay in dilute serum after hydrolysis.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: ug/dL
Arm/Group | Rosiglitazone | Drospirenone/Ethinyl Estradiol | Overweight/Obese Without PCOS | Lean Without PCOS
Number analyzed (Participants) | 17 | 20 | 0 | 0
ug/dL
  DHEAS, Baseline | 165.4 (17.0) | 212.2 (25.4) |  |
  DHEAS, 6 months | 160.9 (17.9) | 197.5 (25.6) |  |

10. Secondary Outcome: Delta Androstenedione at Baseline and 6 Months
Description: Delta Androstenedione was measured by HPLC-tandem mass spectroscopy.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: ng/dL
Arm/Group | Rosiglitazone | Drospirenone/Ethinyl Estradiol | Overweight/Obese Without PCOS | Lean Without PCOS
Number analyzed (Participants) | 17 | 20 | 0 | 0
ng/dL
  Delta Androstenedione, Baseline | 79.2 (11.5) | 82.6 (10.6) |  |
  Delta Androstenedione, 6 months | 58.4 (9.5) | 117.0 (18.2) |  |

11. Secondary Outcome: Delta DHEA at Baseline and 6 Months
Description: Delta DHEA was measured by HPLC-tandem mass spectroscopy.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: ug/dL
Arm/Group | Rosiglitazone | Drospirenone/Ethinyl Estradiol | Overweight/Obese Without PCOS | Lean Without PCOS
Number analyzed (Participants) | 17 | 20 | 0 | 0
ug/dL
  Delta DHEA, Baseline | 817.4 (119.5) | 1001.6 (183.1) |  |
  Delta DHEA, 6 months | 643.4 (102.4) | 1092.1 (188.4) |  |

12. Secondary Outcome: Delta 17-OHProg at Baseline and 6 Months
Description: Delta 17-OHProg (17-hydroxyprogesterone) was measured by HPLC-tandem mass spectroscopy.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: ng/dL
Arm/Group | Rosiglitazone | Drospirenone/Ethinyl Estradiol | Overweight/Obese Without PCOS | Lean Without PCOS
Number analyzed (Participants) | 17 | 20 | 0 | 0
ng/dL
  Delta 17-OHProg, Baseline | 207.0 (37.4) | 169.8 (37.3) |  |
  Delta 17-OHProg, 6 months | 178.0 (49.1) | 175.4 (46.5) |  |

13. Secondary Outcome: Delta 17-OHPreg at Baseline and 6 Months
Description: Delta 17-OHPreg (17-hydroxypregnenolone) was measured by HPLC-tandem mass spectroscopy.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: ng/dL
Arm/Group | Rosiglitazone | Drospirenone/Ethinyl Estradiol | Overweight/Obese Without PCOS | Lean Without PCOS
Number analyzed (Participants) | 17 | 20 | 0 | 0
ng/dL
  Delta 17-OHPreg, Baseline | 912.8 (92.1) | 1024.3 (114.5) |  |
  Delta 17-OHPreg, 6 months | 914.7 (110.9) | 1088.9 (161.0) |  |

14. Secondary Outcome: Cholesterol at Baseline and 6 Months
Description: Cholesterol was measured using the standards of the Centers for Disease Control and Prevention.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Rosiglitazone | Drospirenone/Ethinyl Estradiol | Overweight/Obese Without PCOS | Lean Without PCOS
Number analyzed (Participants) | 17 | 20 | 0 | 0
mg/dL
  Cholesterol, Baseline | 149.5 (8.1) | 156.5 (6.9) |  |
  Cholesterol, 6 months | 146.2 (7.9) | 185.2 (9.1) |  |

15. Secondary Outcome: HDL at Baseline and 6 Months
Description: HDL (high-density lipoprotein) was measured using the standards of the Centers for Disease Control and Prevention.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Rosiglitazone | Drospirenone/Ethinyl Estradiol | Overweight/Obese Without PCOS | Lean Without PCOS
Number analyzed (Participants) | 17 | 20 | 0 | 0
mg/dL
  HDL, Baseline | 42.7 (3.0) | 40.9 (1.9) |  |
  HDL, 6 months | 46.1 (2.1) | 55.0 (2.8) |  |

16. Secondary Outcome: LDL at Baseline and 6 Months
Description: LDL (low-density lipoprotein) was measured using the standards of the Centers for Disease Control and Prevention.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Rosiglitazone | Drospirenone/Ethinyl Estradiol | Overweight/Obese Without PCOS | Lean Without PCOS
Number analyzed (Participants) | 17 | 20 | 0 | 0
mg/dL
  LDL, Baseline | 85.4 (7.6) | 85.9 (6.2) |  |
  LDL, 6 months | 84.3 (7.5) | 97.7 (7.4) |  |

17. Secondary Outcome: Triglycerides at Baseline and 6 Months
Description: Triglycerides were measured using the standards of the Centers for Disease Control and Prevention.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Rosiglitazone | Drospirenone/Ethinyl Estradiol | Overweight/Obese Without PCOS | Lean Without PCOS
Number analyzed (Participants) | 17 | 20 | 0 | 0
mg/dL
  Triglycerides, Baseline | 106.7 (8.1) | 148.4 (14.8) |  |
  Triglycerides, 6 months | 79.2 (6.3) | 163.5 (14.9) |  |

18. Secondary Outcome: Non-HDL Cholesterol at Baseline and 6 Months
Description: Non-HDL cholesterol was measured using the standards of the Centers for Disease Control and Prevention.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Rosiglitazone | Drospirenone/Ethinyl Estradiol | Overweight/Obese Without PCOS | Lean Without PCOS
Number analyzed (Participants) | 17 | 20 | 0 | 0
mg/dL
  Non-HDL cholesterol, Baseline | 65.3 (2.0) | 70.6 (3.5) |  |
  Non-HDL cholesterol, 6 months | 62.3 (1.9) | 87.6 (4.4) |  |

19. Secondary Outcome: Adiponectin at Baseline and 6 Months
Description: Adiponectin was measured by radioimmunoassay.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: ug/mL
Arm/Group | Rosiglitazone | Drospirenone/Ethinyl Estradiol | Overweight/Obese Without PCOS | Lean Without PCOS
Number analyzed (Participants) | 17 | 20 | 0 | 0
ug/mL
  Adiponectin, Baseline | 6.5 (0.7) | 5.9 (0.4) |  |
  Adiponectin, 6 months | 11.6 (1.2) | 6.7 (0.5) |  |

20. Secondary Outcome: Leptin at Baseline and 6 Months
Description: Leptin was measured by radioimmunoassay.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Rosiglitazone | Drospirenone/Ethinyl Estradiol | Overweight/Obese Without PCOS | Lean Without PCOS
Number analyzed (Participants) | 17 | 20 | 0 | 0
ng/mL
  Leptin, Baseline | 43.8 (4.6) | 40.6 (3.8) |  |
  Leptin, 6 months | 42.7 (4.9) | 46.8 (3.9) |  |

21. Secondary Outcome: Hs-CRP at Baseline and 6 Months
Description: hs-CRP(high-sensitivity C-reactive protein) was measured by COAG-Nephelometry.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | Rosiglitazone | Drospirenone/Ethinyl Estradiol | Overweight/Obese Without PCOS | Lean Without PCOS
Number analyzed (Participants) | 17 | 20 | 0 | 0
mg/L
  hs-CRP, Baseline | 2.1 (0.6) | 1.7 (0.5) |  |
  hs-CRP, 6 months | 2.2 (1.0) | 3.8 (0.7) |  |

22. Secondary Outcome: Morning Blood Pressure at Baseline and 6 Months
Description: Morning blood pressure was measured with an automated sphygmomanometer.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Rosiglitazone | Drospirenone/Ethinyl Estradiol | Overweight/Obese Without PCOS | Lean Without PCOS
Number analyzed (Participants) | 17 | 20 | 0 | 0
mm Hg
  Morning Systolic BP, Baseline | 108.2 (2.6) | 108.5 (3.0) |  |
  Morning Diasytolic BP, Baseline | 58.1 (2.0) | 58.1 (1.7) |  |
  Morning Systolic BP, 6 months | 107.5 (2.7) | 112.2 (2.1) |  |
  Morning Diastolic BP, 6 months | 58.7 (1.2) | 59.5 (1.2) |  |

23. Secondary Outcome: Night Blood Pressure at Baseline and 6 Months
Description: Night blood pressure was measured with an automated sphygmomanometer.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Rosiglitazone | Drospirenone/Ethinyl Estradiol | Overweight/Obese Without PCOS | Lean Without PCOS
Number analyzed (Participants) | 17 | 20 | 0 | 0
mm Hg
  Night Systolic BP, Baseline | 117.5 (2.8) | 112.9 (2.1) |  |
  Night Diastolic BP, Baseline | 63.0 (1.5) | 58.6 (1.6) |  |
  Night Systolic BP, 6 months | 115.2 (2.5) | 116.9 (1.9) |  |
  Night Diastolic BP, 6 months | 61.7 (1.5) | 62.6 (1.1) |  |

ADVERSE EVENTS:
Arm/Group | Rosiglitazone | Drospirenone/Ethinyl Estradiol | Overweight/Obese Without PCOS | Lean Without PCOS
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/20 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/17 | 0/20 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The potential unblinding due to the rapid regulation of withdrawal bleeding which may have influenced the dropout rates;the short duration of treatment in contrast to clinical practice where treatment may be for several years.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No